CLINICAL TRIAL: NCT03480061
Title: Dexmedetomidine to Reduce the Incidence of Persistent Cognitive Dysfunction After Open Cardiac Surgery: A Pilot Randomized Trial
Brief Title: Dexmedetomidine to Reduce the Incidence of POCD After Open Cardiac Surgery
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2018
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Delirium; Postoperative Cognitive Dysfunction; Dexmedetomidine; Cognitive Impairment; Depression
MeSH Terms: conditions — Delirium; Postoperative Cognitive Complications; Cognitive Dysfunction; Depression | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Hydrochloride Group (Active Comparator): Patients will receive a loading dose of 1 μg/kg dexmedetomidine prior to transfer to CVICU over 20 min immediately postoperative, followed by continuous infusion of 0.1- 1.0 μg/kg/h for up to 24 hours or until patient is ready for discharge from CVICU (whichever is earlier).
  Interventions: Drug: Dexmedetomidine Hydrochloride Group
- Standard of Care Group (No Intervention): Standard sedation protocols will be followed at the discretion of the attending physician.

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride Group — Dexmedetomidine will be initiated prior to transfer to the CVICU with loading dose of 1 ug kg-1 over approximately 20 minutes. This will be followed by an infusion at 0.1-1.0 ug kg-1h-1 in CVICU for up to 24 hours from the time DEX infusion started or until the patient is ready for discharge from the CVICU (whichever is earlier).
  Other Names: Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine Hydrochloride Group

SUMMARY:
Anesthesia is a drug induced, reversible, comatose state that facilitates surgery and it is widely assumed that cognition returns to baseline after anesthetics have been eliminated. However, many patients have persistent memory impairment for weeks to months after surgery. Cardiac surgery appears to carry the highest risk of postoperative cognitive dysfunction (POCD). These cognitive deficits are associated with increased mortality, prolonged hospital stay and loss of independence. The investigators propose to investigate the role of Dexmedetomidine (DEX) in preventing long-term POCD after cardiac surgery and enhancing early postoperative recovery. It is anticipated that DEX will be the first effective preventative therapy for POCD, improve patient outcomes, and reduce length of stay and healthcare costs.

DETAILED DESCRIPTION:
Dexmedetomidine (DEX), a highly potent and selective α2-adrenoceptors (α2R) agonist used in clinical practice for sedation, analgesia, and anxiolysis, was recently shown to have beneficial effects on early cognitive changes by reducing delirium in humans.It also reduced memory impairment after surgery and isoflurane anesthesia, both in elderly mice (20-22 months) and in pups exposed to anesthesia in the early postnatal period. Importantly, co-treatment with DEX has been shown to restore learning and memory function in rats exposed to propofol in utero. Therefore, the investigators set out to investigate whether DEX has an effect on cognitive dysfunction months after surgery and whether it accelerates cognitive recovery from anesthesia and surgery.

Participants will be randomized 1:1 in permuted blocks of 4 to 8. The randomization sequence will be computer generated and stratified by 2 factors, planned procedure (CABG/CABG + valve or valve only procedure) and study site (for full multicentre trial).

In hospital outcomes include delirium (assessed twice daily post-operative day (POD) 0-10, death, hemodynamic instability requiring vasopressors, time to extubation, re-intubation (and reason), length of stay (in Cardiovascular Intensive Care Unit and total hospital), POCD, depressive symptoms between POD 4-10, post-operative complications (infection [surgical site, sepsis, pneumonia], myocardial infarction, renal replacement therapy, re-operation, cumulative opioid consumption (to POD 4), in-hospital mortality.

Post-operative outcomes include POCD (3/6/12 months), depression (3/6/12 months), mild cognitive impairment (MCI) at 3/6/12 months (defined as 1-2 standard deviations below age matched controls), persistent surgical site pain at sternotomy/thoracotomy/graft harvest site (Brief Pain Inventory, 3/6/12 months), recovery (3,6, 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Planned CABG (including off-pump) or valve replacement (+/- CABG) via sternotomy/thoracotomy, with initial recovery in the Cardiovascular Intensive Care Unit (CVICU)
* age ≥60

Exclusion Criteria:

* Lack of patient consent
* Pregnant or nursing females
* Pre-operative major cognitive dysfunction (CogState Brief Battery score < 80)
* Aortic arch replacement/re-implantation (Bentalls)
* Allergy/contraindication to dexmedetomidine (untreated 2nd degree type 2 or 3rd degree heart block (pacemaker), cirrhosis, HR < 50 , grade 4 LV, renal failure or on renal replacement therapy)
* Unlikely to comply with study assessments (e.g. no fixed address, cannot complete cognitive tests at the 3, 6, and 12 month timepoints)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-08-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | 12 Months
  Ability to recruit 15% a full trail sample size (90 participants)

SECONDARY OUTCOMES:
Completion of follow-up assessments | 3 months
  Ability to achieve 90% follow-up of administering cognitive assessment 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Choi, MD,MSc,FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Sinziana Avramescu, MD,PhD,FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No